CLINICAL TRIAL: NCT05921422
Title: Cognitive Functioning in Children and Adolescents With Cerebral Palsy
Acronym: CPCog-Youth-DK
Status: Recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Center for Rehabilitation of Brain Injury (Center for Hjerneskade) (Unknown); Aarhus University Hospital (Other); University of Copenhagen (Other)
Responsible Party: Principal Investigator, Camilla Funch Uhre, MSc, PhD, Rigshospitalet, Denmark
Other Study IDs: P-2023-155
Record Dates: First submitted 2023-06-19; First posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — Mental Status and Dementia Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case group: Children and adolescents with cerebral palsy who are 11-15 years old, diagnosed with cerebral palsy (any type), and who attend a Danish mainstream school at time of enrollment
  Interventions: Other: Cognitive assessment
- Control group: Children and adolescents without cerebral palsy in the same age range as case-participants (11-15 years old) and attend Danish mainstream schools.
  Interventions: Other: Cognitive assessment

INTERVENTIONS:
Other: Cognitive assessment — All participants will receive cognitive assessment with a core battery (CPCog) and a supplemental battery.
  The core battery includes standardized tests of general cognitive functioning (intelligence) and visual-spatial abilities, as well as a questionnaire on executive functioning in daily life. The supplemental battery assesses attention, executive functioning, memory, fatigue, and symptoms of mental health issues (including symptoms of anxiety, depression, and attention deficit hyperactivity disorder/ADHD).

SUMMARY:
Background: Cerebral palsy (CP) is characterized by motor impairment but commonly involves more widespread difficulties, including cognitive impairment. However, cognitive impairment in CP - especially of a more subtle nature - is often overlooked, despite being associated with substantial academic, social, and emotional problems. In Denmark, the CP follow-up program (CPOP) includes systematic assessment of physical functions, but cognitive assessment is omitted. Prior to starting school, professionals evaluate the school readiness of children with CP, sometimes including a test of general cognitive functioning. Thereafter, cognitive assessments are rarely offered in mainstream schools (Folkeskolen) and can only be accessed if the difficulties are clearly disabling. Recent studies indicate that cognitive assessment needs to be implemented in the follow-up program for school children. For example, one study found that only 42% of students with CP complete mainstream school in Denmark, and international neurocognitive studies have found global cognitive difficulties (lower IQ) and specific impairments in visuo-spatial functions, executive functions, and processing speed in youth with CP. User organizations in the Nordic countries have called for action in recent years, leading to the development of a proposed cognitive follow-up program for children and adolescents with CP, the CPCog, which has yet to be evaluated and implemented in Denmark. Taken together, prior studies and patient experiences emphasize the need for systematic assessment of cognitive functioning in children and adolescents with CP to document the type and extent of cognitive difficulties, secure qualified intervention, and prevent the development of social and emotional problems.

Objective: The main purpose of this study is to characterize cognitive functioning in children and adolescents with CP in Danish mainstream schools. By documenting the extent and type of cognitive impairment associated with CP, we aim to inform future clinical practice and make recommendations for systematic assessment and intervention.

Method: The study is a cross-sectional study with 100 children and adolescents with CP (11-15 years). Each participant will undergo cognitive assessment with the core battery proposed in the Nordic CPCog protocol, including assessment of general cognitive functioning (intelligence), executive functions, and visuo-motor skills. Additionally, participants will undergo supplemental tests of memory, attention, fatigue, and symptoms of psychopathology. Cognitive assessments will take place at two sites: the Neurocenter for Children and Adolescents, Center for Rehabilitation of Brain Injury, and the Center for Clinical Neuropsychology, Children and Adolescents, Rigshospitalet, Copenhagen, Denmark. The project is carried out in collaboration between the neuropediatric and neuropsychological teams associated with the two sites of assessment, as well as the Center for Cerebral Palsy, Rigshospitalet, Aarhus University Hospital, CPOP, and an external advisory board including leading international CP experts.

Results: The CPCog-Youth-DK study will help characterize the cognitive difficulties associated with CP in children and adolescents in mainstream school, which will guide clinical practice and the development and implementation of systematic cognitive assessment and intervention programs. The cognitive assessment protocol will also be evaluated from the perspectives of children and adolescents with CP, parents, and professionals (e.g., assessors and school personnel) to evaluate whether the protocol is tolerable and helpful. Study results will be published in international, peer-reviewed journals, and will be made publicly available via other relevant platforms (such as the websites for the CP clinic at Rigshospitalet, Center for Rehabilitation of Brain Injury, and the Elsass Foundation). Several of the study investigators are directly involved in the current CP follow-up program in Denmark which will aid the process of turning our research into practice.

ELIGIBILITY:
CASE GROUP:

Inclusion Criteria:

* 11-15 years old
* Diagnosed with CP (irrespective of type and severity)
* Attends a Danish mainstream school at time of enrollment

Exclusion Criteria:

- Does not speak or understand Danish at the level necessary to participate (as evaluated by the research team)

CONTROL GROUP:

Inclusion Criteria:

* 11-15 years old
* Attends a Danish mainstream school at time of enrollment

Exclusion Criteria:

* Does not speak or understand Danish at the level necessary to participate (as evaluated by the research team)
* Diagnosed with CP (irrespective of type and severity), traumatic brain injury or other neurological disorder (e.g., epilepsy)

Ages: 11 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children and adolescents with cerebral palsy and healthy control participants (age range: 11-15 years old).
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Global cognitive functioning (IQ) | At first day of assessment
  General cognitive functioning as measured by the GAI from the Wechsler Intelligence Scale for Children, Fifth Edition (WISC-V)
Visuo-spatial functioning | At first day of assessment
  Score from the Beery-Buktenica Developmental Test of Visual Motor Integration (Beery VMI)
Executive functioning | At first day of assessment
  Cognitive regulation index score from the Behavior Rating Inventory of Executive Function - second edition (BRIEF-2), parent version.

SECONDARY OUTCOMES:
Task switching ability | At second day of assessment
  Number of correct words named on the D-KEFS verbal fluency task, and completion time in seconds on the D-KEFS Trail Making task
Attention | At second day of assessment
  Response sensitivity score (d') on the Test of Variables of Attention (T.O.V.A.)
Verbal memory | At second day of assessment
  Scale scores of selected verbal subtests (Word Selective Reminding; Object Recall) from 6the Test of Memory and Learning, Second edition (TOMAL-2)
Visual memory | At second day of assessment
  Scale scores of selected nonverbal subtests (Abstract Visual Memory; Visual Sequential Memory) from the Test of Memory and Learning, Second Edition (TOMAL-2)
Working memory | At second day of assessment
  Working Memory Index score from the WISC-V

OTHER OUTCOMES:
ADHD symptomatology | At second day of assessment
  Total scores of inattention, hyperactivity, and behavior scales of the ADHD-rs questionnaire
Symptoms of autism spectrum disorder | At second day of assessment
  Index score from the Behavior Assessment System for Children, third edition (BASC-3), parent and child version
Symptoms of emotional behavioral disturbance | At second day of assessment
  Index score from the Behavior Assessment System for Children, third edition (BASC-3), parent and child version
Fatigue | At second day of assessment
  PedsQL MFS score
Adaptive functioning | At second day of assessment
  General Adaptive Composite (GAC) score from the Adaptive Behavior Assessment System, Third Edition (ABAS-3)

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Rigshospitalet, Copenhagen
  - Center for Rehabilitation of Brain Injury (Center for Hjerneskade), Copenhagen

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Uhre CF, Caspersen ID, Lose C, Rackauskaite G, Robotham R, Hoei-Hansen CE. Cognitive functioning in children and adolescents with cerebral palsy: protocol for the Danish CPCog-Youth study. BMC Pediatr. 2024 Dec 27;24(1):836. doi: 10.1186/s12887-024-05305-w. PMID 39725891